CLINICAL TRIAL: NCT03479580
Title: Coronary Artery Disease and Coronary Microvascular Disease in Cardiomyopathies Registry
Acronym: 3CRegistry
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Clinique Belledonne (Unknown); Groupe Hospitalier Mutualiste de Grenoble (Other); Centre Hospitalier Annecy Genevois (Other); Centre Hospitalier Metropole Savoie (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC17.215; 2017-A02064-49 (Other: ID RCB)
Record Dates: First submitted 2018-01-23; First posted 2018-03-27 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Hypertrophic; Ischemic; Restrictive Cardiomyopathy; Dilated Cardiomyopathies
Keywords: Cardiomyopathy; Multimodal imaging; Coronary artery disease; Coronary microvascular disease; Prognosis; Atherosclerosis; Myocardial ischemia
MeSH Terms: conditions — Hypertrophy; Ischemia; Cardiomyopathy, Restrictive; Cardiomyopathy, Dilated; Cardiomyopathies; Coronary Artery Disease; Microvascular Angina; Atherosclerosis; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patients with a cardiomyopathy — Prognostic value of coronary artery disease and microvascular disease in the different types of cardiomyopathies.

SUMMARY:
Long-term prognostic value of macrovascular and microvascular coronary artery stenoses in each type of cardiomyopathy.

DETAILED DESCRIPTION:
Coronary artery imaging techniques have taken a central role in the assessment of cardiovascular (CV) diagnosis over the past two decades. Many patients with a cardiomyopathy are also found to have a bystander coronary artery disease, not responsible for their cardiomyopathy. However, the prognostic value of those bystander coronary artery diseases is not known.

Also, new imaging techniques have been developed to assess coronary microvascular disease, but the prognostic value of these findings is not known.

In this study, the investigators evaluate the incidence and the prognosis of bystander coronary artery disease and microvascular disease in patients with ischemic, hypertrophic, dilated and restrictive cardiomyopathies in 5 French centers.

Coronary angiography, cardiac magnetic resonance (CMR), tomographic coronary artery angiography, single-photon emission computed tomography (SPECT), rest and stress trans-thoracic echocardiography (TTE) results will be recorded.

Macrovascular coronary artery disease is defined by :

* a stenosis > 50 % in coronary angiography confirmed with myocardial ischemia (SPECT, stress echocardiography),
* a stenosis > 70 % (50% if it is the left main coronary artery)
* or a stenosis 30-70 % with a fractional flow reserve (FFR) < 0.8 Microvascular disease is defined by an index of microvascular resistance (IMR) >23 or myocardial perfusion heterogeneity imaging (MPHI) > 4 using SPECT or CMR.

Major adverse cardiovascular events (MACE) will be assessed 1 year, 2 years and 5 years after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic
* Dilated
* Hypertrophic
* Restrictive cardiomyopathy.

Exclusion Criteria:

* Pregnant women
* Breastfeeding women
* Patients under legal protection

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female and Male
Study Population: Patients with a cardiomyopathy
Sampling Method: Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2018-02-08 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events | 5 years
  Composite outcome = rate of cardiovascular death, non-fatal myocardial infarction, need for myocardial revascularization by coronary artery bypass graft (CABG) or percutaneous coronary intervention (PCI) > 3 months after enrollment. During follow up

CONTACTS AND LOCATIONS:
Overall Officials: Gilles BARONE-ROCHETTE, PI, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, La Tronche, France